CLINICAL TRIAL: NCT05100875
Title: Social Skills and Emotion Regulation Training "SSERT" for Trauma in Psychosis: A Pilot Feasibility and Acceptability Study
Brief Title: Social Skills and Emotion Regulation Training "SSERT" for Trauma in Psychosis
Acronym: SSERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Martin Lepage, Clinical professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SSERT
Record Dates: First submitted 2021-07-26; First posted 2021-10-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Psychosis; Trauma; Emotion Regulation
MeSH Terms: conditions — Psychotic Disorders; Wounds and Injuries; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention SSERT (Experimental): The SSERT intervention will take place over 10 weekly individual intervention sessions of 60 minutes. SSERT for trauma history in psychosis will draw inspiration from the Skills Training in Affective and Interpersonal Regulation intervention as well as other CBT and DBT-based interventions for emotion regulation and social skills functioning. Therapists will be provided with a semi-structured manual that can be implemented flexibly to consider participant needs.
  Interventions: Behavioral: Social Skills and Emotion Regulation Training "SSERT"

INTERVENTIONS:
Behavioral: Social Skills and Emotion Regulation Training "SSERT" — The SSERT intervention will broadly consist of the following 10 modules: (1) Introducing the Participant to Treatment; (2-3) Emotional Awareness and Recognition; (4-5) Emotion Regulation and Understanding Emotions in the Context of Psychotic Experiences; (6) Living an Emotionally Engaged Life; (7) Understanding Relationship Patterns in the Context of Psychosis; (8) Changing Undesirable Relationship Patterns; (9) Learning to have agency in Relationships; and (10) Flexibility in Relationships and Transitioning to Trauma-Focused Therapy.

SUMMARY:
This study will investigate if the SSERT (Social Skills and Emotion Regulation Training) intervention is feasible and acceptable in individual with psychotic disorder and a history of trauma.

DETAILED DESCRIPTION:
Many individuals with psychotic disorders experience poor functional outcomes such as lower quality of life, lower levels of education, and lower life expectancy. Comorbid mental disorders, such as posttraumatic stress disorder and related posttraumatic stress symptoms tend to aggravate psychotic symptoms and, as a result, worsen functional outcomes. Further, emotion regulation and interpersonal functioning are generally impaired in individuals with psychotic disorders and histories of childhood trauma, and preliminary evidence suggests that these impairments may mediate the relationship between childhood trauma and psychotic symptom severity. Despite the high levels of trauma observed in psychotic populations, the last decade has seen only a modest increase in the number of trials examining the efficacy of trauma interventions in this population. Further, given the initial distress, destabilization, and increased vulnerability that may occur when first engaging in trauma-focused intervention, it has been argued that in those with psychotic disorders, stabilizing/grounding interventions may be a necessary fist step prior to engagement in trauma therapy. This study will thus assess whether the Social Skills and Emotion Regulation Training (SSERT) for Trauma in Psychosis is feasible and acceptable to offer as a preparatory intervention, and will examine its preliminary effect on emotion regulation, interpersonal functioning, and other functional outcomes. SSERT proposes a single-arm baseline with post-intervention design. We will recruit 20 participants with a psychotic disorder, a history of trauma, and an impairment in interpersonal functioning and/or emotion regulation. The intervention will consist of nine weekly hour-long individual sessions and one final 90-minute session. The feasibility of SSERT will be assessed by examining the profile or safety of the study (including whether there are any adverse events reported), the participant flow (missed sessions, attrition rates, retention/completion rates), and through both standardized and qualitative items assessing therapist feedback. The acceptability of SSERT will be assessed subjectively, specifically though participant responses on therapy satisfaction, therapeutic alliance, and motivation for therapy questionnaires. Qualitative analyses will identify common themes and assess participant comments. We expect that SSERT will be both feasible and acceptable to administer to this population. Any expectations regarding the intervention's effect in improving emotion regulation, interpersonal functioning, and other functional outcomes is exploratory. Overall, SSERT may help people with psychotic disorders to better understand how the experience and effect of trauma impacts their relationships and emotion management. The intervention may also help to improve functional outcomes and relationship quality by teaching emotion regulation and grounding strategies, and through learning to become more engaged and flexible in relationships.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosis of a schizophrenia spectrum or other psychotic disorder including affective psychosis;
* (2) trauma history meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) PTSD criterion A;
* (3) at least a mild impairment in either emotional regulation or interpersonal functioning, identified using predetermined cut-offs of ≤ 2 on the Emotion Regulation Skills Questionnaire or ≥ 1 on the Inventory or Interpersonal Problems-32 ;
* (4) at least 18 years of age;
* (5) clinically stable/taking a stable dose of antipsychotic medication;
* (6) French or English-speaking; and
* (7) with no major physical illness.

Exclusion Criteria:

* (1) history of a medical or neurological condition that can affect cognition, which will be verified via participant self-report;
* (2) current severe substance use disorder; and
* (3) an IQ score below 70, estimated using the Wechsler Abbreviated Scale of Intelligence - Two subtest version (vocabulary, matrix reasoning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Participant completion rate | 10 weeks of the intervention
  Feasibility, percentage of participants to complete at least 50% of sessions
Adverse events | 10 weeks of the intervention
  Feasibility, number of recorded adverse events directly associated with the trial
SSERT Feasibility Questionnaire-Therapist | Completion time 10 minutes
  Feasibility, self-report questionnaire completed by the therapist
Working Alliance Inventory-Short Revised | Completion time 5 minutes
  Acceptability, self-report questionnaire
Client Motivation for Therapy Scale | Completion time 5 minutes
  Acceptability, self-report questionnaire
Client Satisfaction Questionnaire | Completion time 5 minutes
  Acceptability/satisfaction, self-report questionnaire
The Satisfaction with Therapy Questionnaire | Completion time 5 minutes
  Acceptability/satisfaction, self-report questionnaire

SECONDARY OUTCOMES:
Emotion Regulation Skills Questionnaire | Completion time 5 minutes
  Emotion regulation, self-report questionnaire
Inventory of Interpersonal Problems- 32 | Completion time 5 minutes
  Interpersonal functioning, self-report questionnaire

OTHER OUTCOMES:
The PTSD Checklist for DSM-5 | Completion time 10 minutes
  Posttraumatic stress symptoms, self-report questionnaire
The Dissociative Experiences Scale II | Completion time 10 minutes
  Dissociative symptoms, self-report questionnaire
Positive and Negative Syndrome Scale-6 (PANSS-6) | Evaluation time 20 minutes
  Psychotic symptoms, observer-rated measure
Psychotic Symptoms Rating Scales, distress dimension | Evaluation time 10 minutes
  Distress associated with psychotic symptoms, observer-rated measure
Beck Cognitive Insight Scale | Completion time 5 minutes
  Metacognition, self-report questionnaire
Overall Anxiety and Severity Impairment Scale | Completion time 5 minutes
  Anxiety, self-report questionnaire
Patient Health Questionnaire-9 | Completion time 5 minutes
  Depression, self-report questionnaire
Brief COPE scale | Completion time 5 minutes
  Coping, self-report questionnaire
Abbreviated- Quality of Life Enjoyment and Satisfaction Questionnaire | Completion time 5 minutes
  Quality of life, self-report questionnaire
Self-Esteem Rating Scale- Short Form | Completion time 5 minutes
  Self-esteem, self-report questionnaire
The Warwick-Edinburgh Mental Well-being Scale | Completion time 5 minutes
  Wellbeing, self-report questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Research Center, Verdun, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No